CLINICAL TRIAL: NCT04988984
Title: Development of Device Kit for Rapid and Sensitive Diagnostic Method for the Tuberculosis; Using Amine Groups Called HI(Homobifunctional Imidoesters),Negative Charge of the Pathogen and Formed Electrical Bonding to Isolate and Concentrate the Pathogen
Brief Title: Development of Automated Molecular Diagnostic Platform for Tuberculosis Diagnosis (New Assay TB)
Acronym: New Assay TB
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Associate Professor, Asan Medical Center
Other Study IDs: 2020-1745
Record Dates: First submitted 2021-07-19; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Tuberculosis Infection
Keywords: New diagnostic platform,TB
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oral swab,BAL, Pleural fluid,Sputum of agreed Subject
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected TB: Patient suspected of TB undergoing diagnostic testing.

SUMMARY:
It is intended for patients who have been admitted to the outpatient or emergency room or are hospitalized For patients who diagnose pulmonary tuberculosis or extrapulmonary tuberculosis using Xpert TB/RIF, additionally, diagnose pulmonary tuberculosis or extrapulmonary tuberculosis using a new diagnostic method, and check the test results. Check whether the tuberculosis bacteria were actually cultured in the sample in the future, and compare the sensitivity and specificity in each test.

Validation in animal model In an animal model (rat) with chronic obstructive pulmonary disease that shows similar characteristics to tuberculosis destructive lung, It will be investigated whether the HI method can be validated by separating and concentrating microbiome for various pathogens including Mycobacterium tuberculosis using HI method. Confirm.

DETAILED DESCRIPTION:
Usefulness of Pulmonary Tuberculosis Diagnosis A comparison of the new diagnostic method with the Xpert TB/RIF test, which is widely used in clinical practice, that can quickly diagnose pulmonary tuberculosis within 1-2 days. ; Considering the sensitivity of the Xpert TB/RIF test as 70% and the sensitivity of the new diagnostic method as 90%, the number of patients with pulmonary tuberculosis required to confirm that the new diagnostic method is useful is estimated as 90 (study power 90%, alpha error = 0.05). And, if 200 patients with suspected pulmonary tuberculosis are registered, it is possible to verify the clinical usefulness compared to Xpert TB/RIF even in 60 AFB smear negative patients. In addition, for the same reason, if 150 additional patients who underwent bronchoscopy were enrolled, it would be possible to compare the diagnosis rate and utility of sputum and bronchoscopy fluid. Waiting for the tuberculosis bacteria culture test for 6 weeks and using the final culture-positive patient as a gold standard for tuberculosis diagnosis -Usefulness of extrapulmonary tuberculosis diagnosis

Millet tuberculosis is disseminated tuberculosis through blood, and there are numerous millet-like lesions in the lungs, but in fact, the positive rate of AFB smear is low due to paucibacillary TB. It is planned to prove the usefulness of the new test method in 35 people with millet tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary TB
* Extrapulmonary TB

Exclusion Criteria:

* under 19

Ages: 19 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 400
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity when using Xpert TB/RIF tests with | From date of experiment until the date of first documented progression assessed upto 100 months
  Comparison of sensitivity and specificity of existing Xpert TB/RIF tests and new diagnostic methods using Homobifunctional Imidoesters (HI) compounds in diagnosing suspected cases of pulmonary tuberculosis and pulmonary tuberculosis
  And the sensitivity and specificity of these two test results are evaluated by waiting for the tuberculosis bacillus culture test for 6 weeks and using the final culture-positive patient as a gold standard for tuberculosis diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Seiwon Lee, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea

REFERENCES:
- [Background] Park YS, Hong SJ, Boo YK, Hwang ES, Kim HJ, Cho SH, Na KI, Cho EH, Shin SS. The national status of tuberculosis using nationwide medical records survey of patients with tuberculosis in Korea. Tuberc Respir Dis (Seoul). 2012 Jul;73(1):48-55. doi: 10.4046/trd.2012.73.1.48. Epub 2012 Jul 31. PMID 23101024
- [Background] Diagnostic Standards and Classification of Tuberculosis in Adults and Children. This official statement of the American Thoracic Society and the Centers for Disease Control and Prevention was adopted by the ATS Board of Directors, July 1999. This statement was endorsed by the Council of the Infectious Disease Society of America, September 1999. Am J Respir Crit Care Med. 2000 Apr;161(4 Pt 1):1376-95. doi: 10.1164/ajrccm.161.4.16141. No abstract available. PMID 10764337
- [Background] Lee JY. Diagnosis and treatment of extrapulmonary tuberculosis. Tuberc Respir Dis (Seoul). 2015 Apr;78(2):47-55. doi: 10.4046/trd.2015.78.2.47. Epub 2015 Apr 2. PMID 25861336
- [Background] Wilkinson RJ, Rohlwink U, Misra UK, van Crevel R, Mai NTH, Dooley KE, Caws M, Figaji A, Savic R, Solomons R, Thwaites GE; Tuberculous Meningitis International Research Consortium. Tuberculous meningitis. Nat Rev Neurol. 2017 Oct;13(10):581-598. doi: 10.1038/nrneurol.2017.120. Epub 2017 Sep 8. PMID 28884751
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Rufai SB, Singh A, Singh J, Kumar P, Sankar MM, Singh S; TB Research Team. Diagnostic usefulness of Xpert MTB/RIF assay for detection of tuberculous meningitis using cerebrospinal fluid. J Infect. 2017 Aug;75(2):125-131. doi: 10.1016/j.jinf.2017.04.010. Epub 2017 May 10. PMID 28501491